CLINICAL TRIAL: NCT06402461
Title: A Randomized Controlled Study Comparing the Effect of Preferential and Random Allocation to Type of Mindfulness Practice in the General Population.
Brief Title: Comparing Random Allocation and Allocation by Preference to Mindfulness Practice
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DClinPsychol2022BobbieScott/1
Record Dates: First submitted 2024-04-29; First posted 2024-05-07 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: 3x2x3: 'group' (preference vs. randomly allocation) by 'practice type' (mindfulness of the breath vs. mindfulness of sounds) by 'time' (baseline vs. post-allocation vs. post-intervention).
Who Masked: Outcomes Assessor
Masking Description: Outcome measures will be collected online using Qualtrics without involvement of a researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Allocation by preference (Experimental): Participants are allocated to the one of the two mindfulness practices that they would prefer to do, based on a short description.
  Interventions: Behavioral: Mindfulness of the breath; Behavioral: Mindfulness of sounds
- Allocation by random (Experimental): Participants are randomly allocated to one of the two mindfulness practices.
  Interventions: Behavioral: Mindfulness of the breath; Behavioral: Mindfulness of sounds
- Control (Active Comparator): Participants listen to an excerpt from an audiobook for an equivalent length of time to the mindfulness practices.
  Interventions: Behavioral: Audiobook control

INTERVENTIONS:
Behavioral: Mindfulness of the breath — A 10 minute, audio guided, mindfulness of the breath meditation of the sort used in mindfulness-based cognitive therapy
  Arms: Allocation by preference; Allocation by random
Behavioral: Mindfulness of sounds — A 10 minute, audio guided, mindfulness of sounds meditation of the sort used in mindfulness-based cognitive therapy
  Arms: Allocation by preference; Allocation by random
Behavioral: Audiobook control — Listening to a 10 minute extract from an audiobook
  Arms: Control

SUMMARY:
The goal of this randomized controlled study is to examine whether allocation based on preference to one of two brief mindfulness meditation practices (mindfulness of the breath or mindfulness of sounds) influences the potentially beneficial effects of these practices, and influences participants' intention to engage in further mindfulness practice. To the end, members of the general public will be randomly assigned to one of three groups: (1) a group in which they choose which of the two mindfulness practices they do; (2) a group in which they are randomly allocated to do one of the mindfulness practices; and (3) a control group that listens to an audiobook extract. The level of mindfulness of each group will be compared, along with some other outcomes.

DETAILED DESCRIPTION:
The study will be an online administered experimental 3x2x3 design, with between-participant factor group (allocated to mindfulness practice based on preference vs. randomly allocated to mindfulness practice vs. audiobook control); a between-participant factor of practice type (mindfulness of the breath vs. mindfulness of sounds), which will be a dummy variable for the control group; and a within-participant factor of time (baseline vs. post-allocation vs. post-intervention). Participants in the 'preference group' will choose which of two mindfulness meditation practices (mindfulness of the breath or mindfulness of sounds) to undertake based on a brief description. Participants in the 'random allocation' group will be allocated to one of the two mindfulness practices at random, and participants in the control group will listen to an excerpt from an audiobook of an equivalent length of time. The primary outcome, state mindfulness, will be measured at all three time-points, as will positive and negative mood. Practice quality and intentional to engage in future mindfulness practice will be measured at post-intervention only.

The following hypotheses will be tested:

H1: Both the allocation by preference and random allocation groups will show greater improvement than the control group on both the primary outcome (baseline to post-intervention change in state mindfulness) and all the secondary outcomes, with the exception of practice quality (which is not applicable for the control group).

H2: The allocation by preference group will show better primary and secondary outcomes than the allocation by random group.

H3: The difference between each mindfulness-practice group and the control group in baseline to post-intervention improvement in mood state will be statistically mediated by baseline to post-intervention increase in state mindfulness.

H4:The difference between the allocation by preference and random allocation groups in baseline to post-intervention change in mood state will be serially, statistically mediated by practice quality and baseline to post-intervention change in state mindfulness respectively, such that participants allocated to the preference group will show higher practice quality, which in turn will statistically predict greater improvement in mindfulness, which in turn will statistically predict greater improvement in mood state.

H5: The same statistical mediation effects as described in H4 above will be observed when the outcome is self-reported intention to practice mindfulness in future, instead of mood state.

ELIGIBILITY:
Inclusion Criteria:

-Resident in the UK

Exclusion Criteria:

* Currently practicing mindfulness meditation more than once per week.
* Experiencing significant mental health problems.
* Believe that practicing mindfulness could cause significant distress.
* Previously practicing mindfulness has caused significant distress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline (T0) to post-intervention (T2) on the Toronto Mindfulness Scale, State Version (TMS-SV; Lau et al., 2006). | Post-intervention (T2; estimated to be on average 20 minutes after baseline)
  The TMS-SV measures two facets of state mindfulness, namely curiosity (on a 0 to 24 scale) and decentering (on a 0 to 28 scale), with higher scores indicating greater state mindfulness.

SECONDARY OUTCOMES:
Change from baseline (T0) to post-allocation (T1) on the Toronto Mindfulness Scale, State Version (TMS-SV; Lau et al., 2006). | Post-allocation (T1; estimated to be on average 5 minutes after baseline)
  As above
Practice Quality-Mindfulness (PQ-M; Del Re et al., 2022) at post-intervention (T2), for the mindfulness practice groups only. | Post-intervention (T2; estimated to be on average 20 minutes after baseline)
  The PQ-M produces two scores (perseverance and receptivity), each ranging from 0 to 100, that measure two aspects of mindfulness practice quality. Higher scores indicate greater quality of mindfulness practice.
Intention to practice mindfulness in future. | Post-intervention (T2; estimated to be on average 20 minutes after baseline)
  Participants will be asked a bespoke question to measure how strong their intention is to practice mindfulness in future, on a scale of 0 to 10, with higher scores indicating greater intention to practice.
Change from baseline (T0) to post-allocation (T1) on the Positive and Negative Affect Schedule - Postive Affect subscale (PANAS-P; Watson et al., 1988) | Post-allocation (T1; estimated to be on average 5 minutes after baseline)
  The PANAS-P measures state positive affect on a 1 to 50 scale, with higher scores indicating greater positive affect.
Change from baseline (T0) to post-intervention (T2) on the Positive and Negative Affect Schedule - Postive Affect subscale (PANAS-P; Watson et al., 1988) | Post-intervention (T2; estimated to be on average 20 minutes after baseline)
  As above
Change from baseline (T0) to post-allocation (T1) on the Positive and Negative Affect Schedule - Negative Affect subscale (PANAS-N; Watson et al., 1988) | Post-allocation (T1; estimated to be on average 5 minutes after baseline)
  The PANAS-N measures state negative affect on a 1 to 50 scale, with higher scores indicating greater negative affect.
Change from baseline (T0) to post-intervention (T2) on the Positive and Negative Affect Schedule - Negative Affect subscale (PANAS-N; Watson et al., 1988) | Post-allocation (T2; estimated to be on average 20 minutes after baseline)
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Bobbie Scott, MSc, Principal Investigator — Canterbury Christ Church University; Fergal Jones, PhD, Study Chair — Canterbury Christ Church University; Sarah Strohmaier, PhD, Study Director — Victoria University, Melbourne
Locations (1):
- Salomons Institute for Applied Psychology, Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Once the study findings have been published, anonymised IPD will be made available to other researchers upon request and/or published via a university repository.
Time Frame: Post-publication for 10 years.
Access Criteria: Data will be made available to researchers or others with legitimate interest (e.g. clinicians and mindfulness teachers).